CLINICAL TRIAL: NCT01483157
Title: Effects of Strength Training With Vascular Occlusion in Patients With Rheumatoid Arthritis: A Randomized Clinical Trial
Brief Title: Vascular Occlusion and Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vascular occlusion and RA
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- low intensity with vascular occlusion (Experimental)
  Interventions: Other: vascular occlusion with exercise trainig
- high intensity resistance training (Experimental)
  Interventions: Other: high intensity resistance training
- no exercise training (No Intervention)

INTERVENTIONS:
Other: vascular occlusion with exercise trainig — twelve weeks of resistance training with vascular occlusion twice a week
  Arms: low intensity with vascular occlusion
Other: high intensity resistance training — twelve weeks of resistance training twice a week
  Arms: high intensity resistance training

SUMMARY:
Resistance exercise plus vascular occlusion may induce greater improvements in strength and muscle mass resistance training alone. The investigators speculate this training strategy could be beneficial in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* female with rheumatoid arthritis
* Disease activity scores > 2.6
* use of anti-TNF-alpha drugs for at least 8 weeks

Exclusion Criteria:

* BMD < 20 kg/m2
* fibromyalgia
* cardiovascular disease

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
muscle strength | twelve weeks

SECONDARY OUTCOMES:
quality of life | twelve weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo - School of Medicine - Clinical Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Rodrigues R, Ferraz RB, Kurimori CO, Guedes LK, Lima FR, de Sa-Pinto AL, Gualano B, Roschel H. Low-Load Resistance Training With Blood-Flow Restriction in Relation to Muscle Function, Mass, and Functionality in Women With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2020 Jun;72(6):787-797. doi: 10.1002/acr.23911. Epub 2020 May 14. PMID 31033228